CLINICAL TRIAL: NCT04142749
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Oltipraz
Brief Title: Oltipraz for Liver Fat Reduction in Patients With Non-alcoholic Fatty Liver Disease Except for Liver Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMK-N01GI1-P3
Record Dates: First submitted 2019-09-19; First posted 2019-10-29 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — oltipraz

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oltipraz (Active Comparator): Oltipraz 30mg
  Interventions: Drug: Oltipraz
- Placebo (Placebo Comparator): Placebo 30mg
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Oltipraz — Total 90mg, By mouth, TID
  Arms: Oltipraz
Drug: Placebos — Total 90mg, By mouth, TID
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Oltipraz inhibits fatty acid synthesis through AMPK-S6K1 pathway and LXRg-SREBP-1c pathway in liver.

DETAILED DESCRIPTION:
Dithiolethiones, a novel class of adenosine monophosphate-activated protein kinase (AMPK) activators, prevent insulin resistance through AMPK-dependent p70 ribosomal S6 kinase-1 (S6K1) inhibition. And it is well known that the modulation of S6K1 by oltipraz inhibited the development of insulin resistance and hyperglycemia through the AMPK-S6K1 pathway.Also some research reported that LXRg (a member of the nuclear hormone receptor)-mediated increases in SREBP-1c (the sterol regulatory element-binding protein-1c gene) promote the expression of lipogenic genes and enhance fatty acid synthesis and oltipraz inhibits LXRg and SREBP-c. Therefore, Oltipraz inhibits fatty acid synthesis through AMPK-S6K1 pathway and LXRg-SREBP-1c pathway in liver.

ELIGIBILITY:
Inclusion Criteria:

* A person the ages of 19 and 75 years old
* Patients with non-alcoholic fatty liver disease other than cirrhosis that meets all of the following criteria:

  1. Abdominal ultrasonography of Screening indicates that the liver is brighter than the spleen or kidneys, causing suspected fatty liver
  2. Persons with liver fat content is 20% or more on the MRS
  3. Those who do not have significant alcohol intake within two years before screening (men: no more than 210 g per week; women: no more than 140 g per week)
  4. Those who with an alcohol use disorder identification test (AUDIT) result point is no more than 7, during screening.
* Persons with body mass index (BMI) more than 23 kg/m2 during screening
* A person who satisfies the following laboratory test results when screening

  1. Platelet ≥ 130,000/㎣
  2. White blood cell (WBC) ≥ 3,000/㎣
  3. Absolute neutrophil count (ANC) ≥ 1,500/㎣
  4. Albumin ≥ 3.5 g/dL
  5. Serum creatinine ≤ 1.5 X upper limit of normal (ULN)
  6. ULN < Alanine transaminase (ALT) or aspartate transaminase (AST) ≤ 250 IU/L
* A person who is willing to maintain the same lifestyle (exercise, alcohol intake, diet, etc.) maintained for at least four weeks before screening during the clinical trial period.
* A person who voluntarily agrees to participate in this clinical trial

Exclusion Criteria:

* A person who has history of following disease or surgery

  1. Malignant tumour with liver cancer
  2. Malignant tumor excluding liver cancer, However, registration is possible in the following cases

     1. If the investigator determines that the patient has been completely cured after maintaining the condition for at least five years
     2. In case of basal cell or squamous cell carcinoma of the skin, the patient is able to maintain a complete condition for more than three years in the case of cainoma in the cervix (CIN) and carcinema in situ (CIS), and other areas.
  3. autoimmune disease (e.g., inflammatory bowel disease, autoimmune hemolytic disease, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, rheumatoid arthritis, severe psoriasis, etc.)
  4. Bariatric surgery within 24 weeks before screening
* A Person who has comorbidity of the following diseases at the time of screening

  1. Liver cirrhosis identified by an epidemiological or histological examination
  2. Cumulative disease (e.g., alcohol liver disease, toxic hepatitis, autoimmune liver disease, metabolic liver disease, biliary closure, etc.) that may indicates liver abnormalities other than non-alcoholic fatty liver disease
  3. A Person who has been infected or has Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV).
  4. Type 1 diabetes or type 2 diabetes (hemoglobin A1c (HbA1c) > 9%)
  5. A person who has positive result of Human immunodeficiency virus antibody (HIV Ab).
  6. A persons with conditions that may affect the effectiveness and safety by investigator
* A person with AST/ALT ratio of more than 2 at screening
* The person who has the following medication history

  1. Persons administered vitamin E (≥ 800 IU/day) or thiazolidatedione drugs or glucagon-like peptide-1 (GLP-1) agonist drugs within 12 weeks prior to screening
  2. Persons who were given antiobestic drug within 12 weeks of screening For example; antiobestic drug with Central nervous system action: Amfepramone, bupropion and naltrexone, cathine, clobenzorex, dexfenfluramine, ephedrine combinations, etilamfetamine, fenfluramine, lorcaserin, mazindol, mefenorex, phentermine, sibutramine, Peripheral neurotic Obesity drugs: Orlistat, Rimonabant, etc
  3. A person who received medications that could cause fatty liver disease within 8 weeks prior to screening For example; Administration of systemic glucocorticoids for more than two weeks Anabolic steroid-based drug, Estrogen-based drug, Azole-based antimicrobial agent, Nucleoside, Nucleotide reverse transcriptase inhibitor-based drug, Tetracycline-based drug, Amiodarone, tamoxifen, methotrexate, valproic acid, etc
  4. A person who administered drugs that may affect the progress of non-alcoholic fatty liver disease within 4 weeks prior to screening or who require administration during clinical trials For example; Silymarin, biphenyl dimethyl dicarboxylate (DDB), ursodeoxycholic acid (UDCA), S-adenosyl-L-methionine (SAMe), betaine, pentoxyfylline, sodium-glucose cotransporter-2 (SGLT-2) inhibitor, omega 3 fatty acid, etc.

     1. However, the following drugs can be registered if they are under stable dosage for at least 12 weeks and are expected to remain unchanged during clinical trials; Sulfonylurea-based drug, metformin, insulin, dipeptidyl peptidase-4 inhibitor (DPP-4 inhibitor), a-glucosidase inhibitor (a-GI), meglitinide-based drug, statin-based drug, fibrate-based drug, nicotinic acid, ezetimibe, beta-blockers based drug, thiazide based drug
* A person who receive non-drug treatment that may affect the liver within 4 weeks prior to screening.
* A person who administered/treated with other clinical trials/medical devices within 4 weeks prior to screening
* Those who are not able to MRS(I)
* A female who is pregnant, may be pregnant, or is lactating
* A person who is not willing to use appropriate contraceptives during this clinical trial.
* A person who is hypersensitive to the Investigational Product
* A person who is deemed ineligible for clinical trials by the investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Variation of liver fat assessed | 24 weeks compared to the baseline
  Variation of liver fat assessed by MRS at 24 weeks compared to the baseline (%)

SECONDARY OUTCOMES:
The variation in the amount of liver fat | 24 weeks compared to the baseline
  The variation in the amount of liver fat assessed by the MRS at the time of 24 weeks compared to the baseline
Variation of liver fat certificate grade | 24 weeks compared to the baseline
  Variation of liver fat certificate grade assessed by ultrasonic waves
Variation of NFS variation | 24 weeks compared to the baseline
  Variation of NFS at 24 weeks compared to the baseline
Variation of liver elasticities and fatty acids | 24 weeks compared to the baseline
  Variation of liver elasticities and fatty acids assessed by fibroscan at 24 weeks time compared to baseline
FIB-4 | 8 weeks, 16 weeks and 24 weeks
  Variation of FIB-4 from 8 weeks, 16 weeks and 24 weeks to baseline
BMI | 8 weeks, 16 weeks and 24 weeks
  BMI variation at 8 weeks, 16 weeks and 24 weeks relative to the baseline
Variation of ALT, AST, γ-glutamyl transferase (GGT) | 8 weeks, 16 weeks and 24 weeks
  Variation of ALT, AST, γ-glutamyl transferase (GGT) in time of 8 weeks, 16 weeks and 24 weeks relative to the baseline
Cholesterol (total, low-density lipoprotein (LDL), high-density lipoprotein (HDL), very low-density lipoprotein (VLDL), triglyceride (TG) | 8 weeks, 16 weeks and 24 weeks
  Variation of Cholesterol (total, low-density lipoprotein (LDL), high-density lipoprotein (HDL), very low-density lipoprotein (VLDL), triglyceride (TG)
Variation of Homeostatic model adjustment-insulin resistance (HOMA-IR) index | 24 weeks compared to the baseline
  Variation of Homeostatic model adjustment-insulin resistance (HOMA-IR = fasting insulin (μU/mL) × fasting glucose (mmol/L) / 22.5)
Waist circumference | 24 weeks compared to the baseline
  The variation of waist circumference compared to the baseline at 24 weeks

OTHER OUTCOMES:
The Variation of biomarkers | 8 weeks, 16 weeks and 24 weeks
  Adipokine (leptin, adiponectin, resistin, TNF-α, IL-6)
The Variation of biomarkers | 8 weeks, 16 weeks and 24 weeks
  CK-18 (M30, M65)
The Variation of biomarkers | 8 weeks, 16 weeks and 24 weeks
  Hepcidine
Variation of liver fat assessed as tissue samples acquired by liver biopsy | 24 weeks compared to the baseline
  Variation of liver fat assessed as tissue samples acquired by liver biopsy at 24 weeks compared to the baseline
Variation of Steatosis assessed as tissue samples acquired by liver biopsy | 24 weeks compared to the baseline
  Variation of Steatosis at 24 weeks compared to the baseline
Variation of lobular inflammation assessed as tissue samples acquired by liver biopsy | 24 weeks compared to the baseline
  Variation of lobular inflammation at 24 weeks compared to the baseline
Variation of ballooning assessed as tissue samples acquired by liver biopsy | 24 weeks compared to the baseline
  Variation of ballooning at 24 weeks compared to the baseline
NAFLD activity scores (NAS) | 24 weeks compared to the baseline
  Variation of NAFLD activity scores (NAS) at 24 weeks compared to the baseline
Correlation between MRS and ultrasound, fibroscan, FIB-4, and biopsy results | 24 weeks compared to the baseline
  Correlation between MRS and ultrasound, fibroscan, FIB-4, and biopsy results

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Jun Kim, MD.PhD, Principal Investigator — Seoul Nat'l Uni. Hospital; Changuk Kim, MD.PhD, Principal Investigator — The Catholic University of Korea, Uijeongbu ST. Mary's Hospital; Gapjin Chun, MD.PhD, Principal Investigator — Gangneung Asan Medical Center; Taehui Lee, MD.PhD, Principal Investigator — Kunyang University Hospital; Byeongguk Jang, MD.PhD, Principal Investigator — Keimyung University Dongsan Medical Center; Yanghyeon Baek, MD.PhD, Principal Investigator — Dong-A University Hospital; Byeonggwan Kim, MD.PhD, Principal Investigator — Boramae Hospital; Yeongseok Kim, MD.PhD, Principal Investigator — Soonchunhyang University Hospital; Jaeyeong Chang, MD.PhD, Principal Investigator — Soonchunhyang University Hospital; Jaeyeong Jung, MD.PhD, Principal Investigator — Ajou University School of Medicine; Hyeonung Lee, MD.PhD, Principal Investigator — Yonsei University Gangnam Severance Hospital; Doyeong Kim, MD.PhD, Principal Investigator — Severance Hospital; Munyeong Kim, MD.PhD, Principal Investigator — Wonju Severance Christian Hospital; Junseong Lee, MD.PhD, Principal Investigator — Inje University Ilsan Baek Hospital; Jinu Lee, MD.PhD, Principal Investigator — Inha University Hospital; Hyeongjun Kim, MD.PhD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Sanghun Park, MD.PhD, Principal Investigator — Hallym University Gangnam Sungsim Hospital; Daewon Jun, MD.PhD, Principal Investigator — Hanyang University; Chun Kyun Lee, MD.PhD, Principal Investigator — National Health Insurance Service Ilsan Hospital; Jaeyun Jung, MD.PhD, Principal Investigator — National medical center; Jihun Kim, MD.PhD, Principal Investigator — Korea University Guro Hospital; Huieon Kim, MD.PhD, Principal Investigator — Catholic University Bucheon ST. Mary's Hospital
Locations (21):
- South Korea (21):
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital, Uijeongbu-si, Gyeonggi-do
  - Inha University Hospital, Incheon, Junggu
  - Catholic University Bucheon ST. Mary's Hospital, Bucheon-si
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Gangneung Asan Medical Center, Gangneung-si
  - NHUS Ilsan Hospital, Goyang-si
  - Seoul National University Hospital, Seoul
  - Boramae Hospital, Seoul
  - Chung-Ang University Hosptial, Seoul
  - Hallym University Gangnam Sungsim Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - National Medical Center, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Yonsei University Gangnam Severance Hospital, Seoul
  - Ajou University School of Medicine, Suwon
  - Wonju Severance Christian Hospital, Wanju